CLINICAL TRIAL: NCT02653521
Title: The Clinical Physics Research of Image Guided Adaptive Radiation Therapy for Esophagus Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Deng Xiaowu, Director of radiotherapy department, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M201505
Record Dates: First submitted 2015-12-28; First posted 2016-01-12 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Adaptive Radiation Therapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- adaptive radiation therapy (ART) (Experimental): 40 patients treated with ART, using dose adaptation method to match the change of PTV and movement of OARs and achieve an optimal dose distribution using online CBCT images.
  Interventions: Radiation: Dose adaptation
- the control group (No Intervention): 40 patients treated with original plan for full treatment course.

INTERVENTIONS:
Radiation: Dose adaptation — Replanning the treatment to adapt the change of PTV and movement of OARs to achieve an optimal dose distribution using online CBCT images.
  Arms: adaptive radiation therapy (ART)

SUMMARY:
The purpose of this study is to evaluate the benefit of adaptive radiation therapy (adaptive radiation therapy, ART) for esophageal cancer, using dose tracking technique with online images and deformable registration.

DETAILED DESCRIPTION:
The aim of study is to evaluate the benefit of adaptive radiation therapy(ART) for esophageal cancer. 80 patients with locally advanced esophageal cancer will be treated with 3D-CRT(three dimensional conformal radiotherapy, 3D-CRT)/IMRT(intensity modulated radiotherapy, IMRT), dividing to experimental group and control group (40 patients each). All patients are kVCT(kilo-voltage computed tomography, kVCT) scanned weekly(the fifth fraction in a week) and CBCT (cone beam computed tomography, CBCT) scanned per fraction before treatment. Irradiated dose distribution of each patient is calculated using the CBCT images corrected with validated modelling and accumulate the volumetric dose for all PTV(planning target volume,PTV) and OARs(organs at risk, OAR) using deformable registration algorithm. For the experimental group, replan the treatment when the target volume is not covered by the prescribed dose or OARs is overdose beyond the action level to achieve an optimal dose distribution. Conversely, no action is taken in the control group and the original plan will be used for the full treatment course. Dosimetric parameters (such as the ratio of target coverage, the mean dose of OARs, etc) ,treatment toxicities (such as radiation pneumonitis and esophagitis), PFS（Progress Free Survival,PFS）and OS（Overall Survival, OS）of the two groups will be analyzed and compared in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with locally advanced esophageal cancer
* ECOG(Eastern Cooperative Oncology Group, ECOG) physical status score：0-2
* Charlson complications index score≤4
* First second forced expiratory volume ≥1 liter
* Patients and their families agreed and signed the informed consent

Exclusion Criteria:

* Previous treatment with other malignant tumor
* Had anti-tumor treatment, including (chemotherapy, radiotherapy, surgery)
* Any taboo disease or condition of radiotherapy and chemotherapy
* With malignant pleural effusion and pericardial effusion
* Participated to other clinical test within 30 days before this experiment
* With uncontrolled seizures or loss of mental self-control
* Drug takers, chronic alcoholism, and HIV/AIDS patients
* Has a history of severe allergic or specific physique
* Researchers think that is unfavorable to the test

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-12-30; Primary Completion 2018-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Toxicity of treatment | One year
  Evaluating the treatment toxicity weekly during treatment course and at the time of one year after treatment according to the NCI CTCAE 4.0 (The National Cancer Institute Common Terminology Criteria for Adverse Events,NCI-CTCAE, Version 4.0).

SECONDARY OUTCOMES:
Progress Free Survival(PFS） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  the length of time during and after the treatment of a disease
Overall Survival（OS） | 2 years
  The survival time from the start of treatment to death or the time of the last follow-up of this study.

OTHER OUTCOMES:
Dosimetric Parameters | Six weeks
  Accumulated dose distribution of the full treatment course.

CONTACTS AND LOCATIONS:
Overall Officials: Deng Xiaowu, PHD., Study Director — Sun Yat-sen University; Liu Hui, PHD., Study Director — Sun Yat-sen University; Peng Yinglin, MD, Principal Investigator — Sun Yat-sen University; Qiu Bo, PHD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hawkins MA, Brooks C, Hansen VN, Aitken A, Tait DM. Cone beam computed tomography-derived adaptive radiotherapy for radical treatment of esophageal cancer. Int J Radiat Oncol Biol Phys. 2010 Jun 1;77(2):378-83. doi: 10.1016/j.ijrobp.2009.05.045. Epub 2009 Sep 21. PMID 19775828
- [Background] Sriram P, Syamkumar SA, Kumar JS, Prabakar S, Dhanabalan R, Vivekanandan N. Adaptive volumetric modulated arc treatment planning for esophageal cancers using cone beam computed tomography. Phys Med. 2012 Oct;28(4):327-32. doi: 10.1016/j.ejmp.2011.10.006. Epub 2011 Nov 10. PMID 22079402